CLINICAL TRIAL: NCT01788670
Title: Hydroxytyrosol as an Endogenous and Natural Antioxidant: Modulation by Alcohol Intake. Substudy 1. Evaluating the Relevance of the Ethanol Dose in the Generation of Endogenous Hydroxytyrosol (DOPET).
Brief Title: Relevance of the Ethanol Dose in the Generation of Endogenous Hydroxytyrosol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fundacion IMIM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Hidroxitirosol/FIS/1
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Contribution of Ethanol on Hydroxytyrosol Formation
Keywords: Antioxidants, Central Nervous System Agents
MeSH Terms: interventions — Ethanol; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Water (Placebo Comparator): Lemon-flavoured water (150 ml)
  Interventions: Other: Water
- Ethanol high dose (Active Comparator): The high dose corresponds to 30 g of ethanol in pilot cohort 1, to 12 g of ethanol in pilot cohort 2 and to 42 g of ethanol in pilot cohort 3. For the definitive study the high dose corresponds to 30 g of ethanol. Ethanol was administered as a single dose of pure ethanol diluted in lemon-flavoured water (150 ml each beverage).
  Interventions: Dietary Supplement: Ethanol
- Ethanol low dose (Active Comparator): The low dose corresponds to 18 g of ethanol in pilot cohort 1, to 6 g of ethanol in pilot cohort 2 and to 24 g of ethanol in pilot cohort 3. For the definitive study the low dose corresponds to 18 g of ethanol. Ethanol was administered as a single dose of pure ethanol diluted in lemon-flavoured water (150 ml each beverage).
  Interventions: Dietary Supplement: Ethanol

INTERVENTIONS:
Dietary Supplement: Ethanol
  Arms: Ethanol high dose; Ethanol low dose
Other: Water
  Arms: Water

SUMMARY:
Health benefits for humans derived from low dose intake of ethanol could partially be explained by its interaction with dopamine (DA) oxidative metabolism. Ethanol is expected to induce an increase in the formation of a DA minor metabolite: DOPET (hydroxytyrosol). Hydroxytyrosol is one of the most potent antioxidants present in Mediterranean Diet. The study is aimed at establishing the contribution of ethanol on hydroxytyrosol formation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* The body mass index (BMI=weigh/height2) will range from 19 to 27 kg/m2, and the weight from 50 to 110 kg.
* Understanding and accepting the study procedures and signing the informed consent.

Exclusion Criteria:

* Not meeting the inclusion criteria.
* History or clinical evidence of alcoholism, drug abuse, or regular use of psychoactive drugs.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* History of psychiatric disorders.
* Smokers of more than 20 cigarettes per day.
* Taking more than 30 g of alcohol a day
* Regular use of any drug in the month prior to the study sessions.The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks.
* Subjects with intolerance or adverse reactions to ethanol
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.

To be eligible, the subjects must agree to follow a diet free from ethanol and olive oil in the 72 hours prior to the start of each session and until the end of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Hydroxytyrosol biological fluids concentrations | 0-24h after administration
  Hydroxytyrosol concentrations in plasma and urine

SECONDARY OUTCOMES:
Subjective drunkenness | 0-6h after administration
  Ethanol subjective effects measured using a visual analog scale
Vital signs | 0-6h after administration
  Blood pressure, oral temperature and heart rate
Ethanol concentration | 0-6h after administration
  Ethanol blood concentrations
Ethanol metabolites concentrations | 0-24h after administration
  Ethanol metabolites recovery in urine
Dopamine metabolites concentrations | 0-24h after administration
  Dopamine metabolites recovery in urine

CONTACTS AND LOCATIONS:
Overall Officials: Magí Farré, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Perez-Mana C, Farre M, Pujadas M, Mustata C, Menoyo E, Pastor A, Langohr K, de la Torre R. Ethanol induces hydroxytyrosol formation in humans. Pharmacol Res. 2015 May-Jun;95-96:27-33. doi: 10.1016/j.phrs.2015.02.008. Epub 2015 Mar 20. PMID 25801942